CLINICAL TRIAL: NCT01897766
Title: AN INVESTIGATION INTENDED TO EVALUATE THE LONG-TERM EFFICACY AND SAFETY OF GENOTROPIN IN CHILDREN WITH SGA DWARFISM WITHOUT EPIPHYSEAL CLOSURE. (RETROSPECTIVE STUDY)
Brief Title: Special Investigation Of Genotropin Long Follow-Up For Patients With A Small For Gestational Age "Scoped for Japanese"
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A6281314
Record Dates: First submitted 2013-07-09; First posted 2013-07-12 (Estimated); Results first posted 2020-02-11 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-08

CONDITIONS: Small for Gestational Age (SGA)
Keywords: Genotropin; Somatropin; Long Term Follow-Up; Special Investigation; Small for Gestational Age; SGA
MeSH Terms: interventions — Human Growth Hormone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Somatropin: Patients administered Somatropin.
  Interventions: Drug: Somatropin

INTERVENTIONS:
Drug: Somatropin — 0.23 mg to 0.48 mg/kg/week
  Other Names: Genotropin

SUMMARY:
The objective of this surveillance is to collect Safety and Effectiveness information for Long term Use of Somatropin for Patients with a Small for Gestational Age (SGA).

DETAILED DESCRIPTION:
All the patients whom an investigator prescribes Genotropin should be registered consecutively until the number of subjects reaches target number in order to extract patients enrolled into the investigation at random.

ELIGIBILITY:
Inclusion Criteria:

* A patient who was administered Somatropin (Genotropin).

Exclusion Criteria:

* N/A.

Ages: 2 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: * A patients who is diagnosed for SGA. (SGA is defined as birth weight and/or length at least 2 standard deviations (SDs) below the mean for gestational age (<or=-2 SD)).
  * A patient who is SGA and older than 3 years.
  * A patient who has persistent short stature (i.e., remaining at least 2.5 SD below the mean for chronologic age).
Sampling Method: Probability Sample
Enrollment: 482 (Actual)
Dates: Start 2013-09-05 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6281314&StudyName=Special%20Investigation%20Of%20Genotropin%20Long%20Follow-Up%20For%20Patients%20With%20A%20Small%20For%20Gestational%20Age%20%28SGA%29

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: It is a retrospective study. Data was collected for participants from July 2005 - February 2017(approximately over 11 years 6 months).
Groups:
- Genotropin [Somatropin (Genetical Recombination)]: Participants who received Genotropin treatment in a real world clinic setting as prescribed in clinical practice from July 2005 - February 2017. Data was observed retrospectively.
Period: Overall Study
Arm/Group | Genotropin [Somatropin (Genetical Recombination)]
Started | 482
Completed | 482
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Participants enrolled in this study.
Arm/Group | Genotropin [Somatropin (Genetical Recombination)]
Number analyzed (Participants) | 482
Age, Customized [Number; unit: Participants]
  <5 years | 220
  ≥5 and <7 years | 95
  ≥7 years | 167
Sex/Gender, Customized [Number; unit: Participants]
  Male | 240
  Female | 242
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Drug Reaction (ADR)
Description: An adverse drug reaction (ADR) was any untoward medical occurrence attributed to Genotropin in a participant who received Genotropin. A serious ADR (SADR) was an ADR resulting in any of the following out comes or deemed significant for any other reason: death; life-threatening experience (immediate risk of dying); initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly. Relatedness to Genotropin was assessed by the physician.
Time Frame: Approximately 11.58 years
Population: The safety analysis set comprised of participants who satisfied the inclusion criteria and had received Genotropin.
Measure: Number; unit: Participants
Arm/Group | Genotropin [Somatropin (Genetical Recombination)]
Number analyzed (Participants) | 482
Participants
  ADR | 24
  SADR | 4

2. Primary Outcome: Change in Height Velocity Standard Deviation (SD) Score for Chronological Age From Baseline At Year 1
Description: Change in height Velocity SD score from baseline was calculated. Height Velocity SD score = (Height - Standard height for chronological age of gender) / SD. An SD score indicates how far a participant's score deviates from the mean of the reference population; an SD score higher than the mean gives a positive SD score whereas an SD score lower than the mean gives a negative SD score. SD score indicates how similar participant was to reference population.
Time Frame: Baseline, Year 1
Population: The efficacy analysis set comprised of participants in the safety analysis set who had effectiveness evaluation at least once. Here "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: SD score
Arm/Group | Genotropin [Somatropin (Genetical Recombination)]
Number analyzed (Participants) | 324
SD score | 4.1 (3.06)

3. Primary Outcome: Change in Height Velocity Standard Deviation (SD) Score for Chronological Age From Baseline at Year 2
Description: as for outcome 2
Time Frame: Baseline, Year 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: SD score
Arm/Group | Genotropin [Somatropin (Genetical Recombination)]
Number analyzed (Participants) | 243
SD score | 3.0 (2.92)

4. Primary Outcome: Change in Height Velocity Standard Deviation (SD) Score for Chronological Age From Baseline at Year 3
Description: as for outcome 2
Time Frame: Baseline, Year 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: SD score
Arm/Group | Genotropin [Somatropin (Genetical Recombination)]
Number analyzed (Participants) | 169
SD score | 2.5 (2.53)

5. Primary Outcome: Change in Height Velocity Standard Deviation (SD) Score for Chronological Age From Baseline at Year 4
Description: as for outcome 2
Time Frame: Baseline, Year 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: SD score
Arm/Group | Genotropin [Somatropin (Genetical Recombination)]
Number analyzed (Participants) | 146
SD score | 2.6 (2.81)

6. Primary Outcome: Change in Height Velocity Standard Deviation (SD) Score for Chronological Age From Baseline at Year 5
Description: as for outcome 2
Time Frame: Baseline, Year 5
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: SD score
Arm/Group | Genotropin [Somatropin (Genetical Recombination)]
Number analyzed (Participants) | 137
SD score | 2.3 (2.74)

7. Primary Outcome: Change in Height Velocity Standard Deviation (SD) Score for Chronological Age From Baseline at Year 6
Description: as for outcome 2
Time Frame: Baseline, Year 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: SD score
Arm/Group | Genotropin [Somatropin (Genetical Recombination)]
Number analyzed (Participants) | 101
SD score | 2.4 (3.07)

8. Primary Outcome: Change in Height Velocity Standard Deviation (SD) Score for Chronological Age From Baseline at Year 7
Description: as for outcome 2
Time Frame: Baseline, Year 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: SD score
Arm/Group | Genotropin [Somatropin (Genetical Recombination)]
Number analyzed (Participants) | 51
SD score | 2.4 (3.86)

9. Primary Outcome: Change in Height Velocity Standard Deviation (SD) Score for Chronological Age From Baseline at Year 10
Description: as for outcome 2
Time Frame: Baseline, Year 10
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: SD score
Arm/Group | Genotropin [Somatropin (Genetical Recombination)]
Number analyzed (Participants) | 1
SD score | -1.6 (NA) — Only 1 subject evaluable hence standard deviation could not be estimated.

10. Primary Outcome: Change in Height Standard Deviation (SD) Score for Chronological Age From Baseline at Year 1
Description: Change in height SD score from baseline was calculated. Height SD score = (Height - Standard height for chronological age of gender) / SD. An SD score indicates how far a participant's score deviates from the mean of the reference population; an SD score higher than the mean gives a positive SD score whereas an SD score lower than the mean gives a negative SD score. SD score indicates how similar participant was to reference population.
Time Frame: Baseline, Year 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: SD score
Arm/Group | Genotropin [Somatropin (Genetical Recombination)]
Number analyzed (Participants) | 388
SD score | 0.6 (0.36)

11. Primary Outcome: Change in Height Standard Deviation (SD) Score for Chronological Age From Baseline at Year 2
Description: as for outcome 10
Time Frame: Baseline, Year 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: SD score
Arm/Group | Genotropin [Somatropin (Genetical Recombination)]
Number analyzed (Participants) | 315
SD score | 0.9 (0.49)

12. Primary Outcome: Change in Height Standard Deviation (SD) Score for Chronological Age From Baseline at Year 3
Description: as for outcome 10
Time Frame: Baseline, Year 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: SD score
Arm/Group | Genotropin [Somatropin (Genetical Recombination)]
Number analyzed (Participants) | 233
SD score | 1.1 (0.51)

13. Primary Outcome: Change in Height Standard Deviation (SD) Score for Chronological Age From Baseline at Year 4
Description: as for outcome 10
Time Frame: Baseline, Year 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: SD score
Arm/Group | Genotropin [Somatropin (Genetical Recombination)]
Number analyzed (Participants) | 223
SD score | 1.3 (0.63)

14. Primary Outcome: Change in Height Standard Deviation (SD) Score for Chronological Age From Baseline at Year 5
Description: as for outcome 10
Time Frame: Baseline, Year 5
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: SD score
Arm/Group | Genotropin [Somatropin (Genetical Recombination)]
Number analyzed (Participants) | 205
SD score | 1.3 (0.71)

15. Primary Outcome: Change in Height Standard Deviation (SD) Score for Chronological Age From Baseline at Year 6
Description: as for outcome 10
Time Frame: Baseline, Year 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: SD score
Arm/Group | Genotropin [Somatropin (Genetical Recombination)]
Number analyzed (Participants) | 136
SD score | 1.4 (0.81)

16. Primary Outcome: Change in Height Standard Deviation (SD) Score for Chronological Age From Baseline at Year 7
Description: as for outcome 10
Time Frame: Baseline, Year 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: SD score
Arm/Group | Genotropin [Somatropin (Genetical Recombination)]
Number analyzed (Participants) | 72
SD score | 1.4 (0.87)

17. Primary Outcome: Change in Height Standard Deviation (SD) Score for Chronological Age From Baseline at Year 9
Description: as for outcome 10
Time Frame: Baseline, Year 9
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: SD score
Arm/Group | Genotropin [Somatropin (Genetical Recombination)]
Number analyzed (Participants) | 1
SD score | 2.1 (NA) — Only 1 subject evaluable hence standard deviation could not be estimated.

18. Primary Outcome: Change in Height Standard Deviation (SD) Score for Chronological Age From Baseline at Year 10
Description: as for outcome 10
Time Frame: Baseline, Year 10
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: SD score
Arm/Group | Genotropin [Somatropin (Genetical Recombination)]
Number analyzed (Participants) | 1
SD score | 1.8 (NA) — Only 1 subject evaluable hence standard deviation could not be estimated.

19. Secondary Outcome: Height Standard Deviation (SD) Score at Puberty and at Near Final Height in Participants Who Reached Near Final Height
Description: Height SD score = (Height - Standard height for chronological age of gender) / SD. An SD score indicates how far a participant's score deviates from the mean of the reference population; an SD score higher than the mean gives a positive SD score whereas an SD score lower than the mean gives a negative SD score. SD score indicates how similar participant was to reference population. Near final height was defined as the height at one of the following conditions: the annual height velocity became less than 2 cm/year after reaching the maximum height in puberty, bone age reached 17 years old and older for male and 15 years old and older for female, or the reason for discontinuation was that subject reached the near final height or had epiphyseal closure.
Time Frame: Baseline, At Puberty, At Near Final Height within the span of approximately maximum of 11.58 years
Population: The efficacy analysis set comprised of participants in the safety analysis set who had effectiveness evaluation at least once. Among the efficacy analysis set, the participants who reached near final height was analyzed.
Measure: Mean (Standard Deviation); unit: SD score
Arm/Group | Genotropin [Somatropin (Genetical Recombination)]
Number analyzed (Participants) | 34
SD score
  At baseline: number analyzed (Participants) | 31
  At baseline | -3.1 (0.77)
  At puberty: number analyzed (Participants) | 26
  At puberty | -2.8 (0.86)
  At near final height: number analyzed (Participants) | 32
  At near final height | -2.5 (1.16)

20. Secondary Outcome: Change in Height Standard Deviation (SD) Score at Puberty and at Near Final Height in Participants Who Reached Near Final Height From Baseline
Description: Change in height SD score from baseline was calculated. Height SD score = (Height - Standard height for chronological age of gender) / SD. An SD score indicates how far a participant's score deviates from the mean of the reference population; an SD score higher than the mean gives a positive SD score whereas an SD score lower than the mean gives a negative SD score. SD score indicates how similar participant was to reference population. Near final height was defined as the height at one of the following conditions: the annual height velocity became less than 2 cm/year after reaching the maximum height in puberty, bone age reached 17 years old and older for male and 15 years old and older for female, or the reason for discontinuation was that subject reached the near final height or had epiphyseal closure.
Time Frame: Baseline, At Puberty, At Near Final Height within the span of approximately maximum of 11.58 years
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: SD score
Arm/Group | Genotropin [Somatropin (Genetical Recombination)]
Number analyzed (Participants) | 34
SD score
  Change at At puberty: number analyzed (Participants) | 24
  Change at At puberty | 0.3 (0.36)
  Change At near final height: number analyzed (Participants) | 29
  Change At near final height | 0.6 (0.74)

ADVERSE EVENTS:
Time Frame: Approximately 11.58 years
Description: The frequency of adverse events. The same event may appear as both an adverse event and a serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in one subject and as non-serious in another subject, or one subject may have experienced both serious and non-serious events during the study.
Arm/Group | Genotropin [Somatropin (Genetical Recombination)]
All-Cause Mortality (participants affected / at risk) | 1/482
Serious Adverse Events (participants affected / at risk) | 32/482
Other Adverse Events (participants affected / at risk) | 105/482
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Genotropin [Somatropin (Genetical Recombination)] (N=482)
Acute sinusitis (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 1
Campylobacter gastroenteritis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 2
Meningitis bacterial (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Febrile convulsion (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Cardiac disorder (Cardiac disorders) | 1
Kawasaki's disease (Vascular disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 1
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1
Scoliosis (Musculoskeletal and connective tissue disorders) | 4
Synovial disorder (Musculoskeletal and connective tissue disorders) | 1
Cryptorchism (Congenital, familial and genetic disorders) | 1
Condition aggravated (General disorders) | 2
Patella fracture (Injury, poisoning and procedural complications) | 1
Snake bite (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Genotropin [Somatropin (Genetical Recombination)] (N=482)
Lymphadenitis (Blood and lymphatic system disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Arnold-Chiari malformation (Congenital, familial and genetic disorders) | 1
Spine malformation (Congenital, familial and genetic disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 2
Thyroiditis (Endocrine disorders) | 1
Conjunctivitis allergic (Eye disorders) | 3
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 4
Pigmentation lip (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Injection site haemorrhage (General disorders) | 1
Injection site urticaria (General disorders) | 1
Pyrexia (General disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 5
Food allergy (Immune system disorders) | 1
Seasonal allergy (Immune system disorders) | 1
Adenoviral upper respiratory infection (Infections and infestations) | 1
Beta haemolytic streptococcal infection (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 17
Bronchitis viral (Infections and infestations) | 1
Dermatitis infected (Infections and infestations) | 1
Ear infection (Infections and infestations) | 1
Erythema infectiosum (Infections and infestations) | 1
Exanthema subitum (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 12
H1N1 influenza (Infections and infestations) | 1
Impetigo (Infections and infestations) | 3
Influenza (Infections and infestations) | 14
Molluscum contagiosum (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 4
Oral herpes (Infections and infestations) | 1
Otitis externa (Infections and infestations) | 1
Otitis media (Infections and infestations) | 7
Otitis media acute (Infections and infestations) | 1
Parotitis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 3
Pneumonia (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 1
Streptococcal infection (Infections and infestations) | 2
Subcutaneous abscess (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Tracheobronchitis mycoplasmal (Infections and infestations) | 1
Varicella (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Meniscus injury (Injury, poisoning and procedural complications) | 1
Thermal burn (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 4
Aspartate aminotransferase increased (Investigations) | 2
Blood alkaline phosphatase increased (Investigations) | 1
Blood cholesterol increased (Investigations) | 1
Blood glucose increased (Investigations) | 2
Blood thyroid stimulating hormone decreased (Investigations) | 1
Blood thyroid stimulating hormone increased (Investigations) | 1
Blood urea increased (Investigations) | 1
Blood urine present (Investigations) | 1
Body mass index increased (Investigations) | 1
Glucose urine (Investigations) | 1
Glycosylated haemoglobin increased (Investigations) | 1
Insulin-like growth factor increased (Investigations) | 2
Protein urine present (Investigations) | 1
White blood cell count increased (Investigations) | 1
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 3
Hyperinsulinaemia (Metabolism and nutrition disorders) | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1
Obesity (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Arthropathy (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Scoliosis (Musculoskeletal and connective tissue disorders) | 2
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neurofibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Febrile convulsion (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Orthostatic intolerance (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 5
Autism spectrum disorder (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Tic (Psychiatric disorders) | 1
Orthostatic proteinuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 2
Renal glycosuria (Renal and urinary disorders) | 2
Renal haemorrhage (Renal and urinary disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 8
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 17
Asteatosis (Skin and subcutaneous tissue disorders) | 3
Blister (Skin and subcutaneous tissue disorders) | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 5
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 3
Urticaria (Skin and subcutaneous tissue disorders) | 2
Oral surgery (Surgical and medical procedures) | 1
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2013-07-02): https://cdn.clinicaltrials.gov/large-docs/66/NCT01897766/Prot_000.pdf
  • Statistical Analysis Plan (2016-10-27): https://cdn.clinicaltrials.gov/large-docs/66/NCT01897766/SAP_001.pdf